CLINICAL TRIAL: NCT05113810
Title: A Pilot, Randomized, Open-label Trial to Determine the Feasibility, Safety, Efficacy, and Pharmacokinetics of Nebulized HCQ01for the Treatment of Patients With COVID-19
Brief Title: The Potential Use of Nebulized Hydroxychloroquine for the Treatment of COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ministry of Health Jordan (Other Government)
Collaborators: King Hussein Cancer Center (Other); ACDIMA Biocenter (Other); Amman Pharmaceutical Industries (Unknown); Sana Pharmaceutical Industry (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1093-2021
Record Dates: First submitted 2021-11-06; First posted 2021-11-09 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: 2019 Novel Coronavirus
Keywords: COVID-19; Inhaled/nebulized Hydroxychloroquine
MeSH Terms: conditions — COVID-19; Respiratory Aspiration | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First Arm (Hydroxychloroquine sulfate, 5 days) (Experimental): Participants will receive continued standard of care therapy (SOC) for COVID-19 together with 2 ml HCQ01 (12.5 mg/ml) twice a day for 5 consecutive days.
  Interventions: Drug: HCQ01
- Second Arm (Continued Standard of Care (SOC) Therapy) (Active Comparator): Participants will receive continued standard of care therapy for COVID-19
  Interventions: Other: standard of care (SOC) for COVID-19

INTERVENTIONS:
Drug: HCQ01 — HCQ01 is a sterile, clear and colorless, ready-to-use aqueous nebulizer solution. Hydroxychloroquine sulfate administered via nebulization
  Arms: First Arm (Hydroxychloroquine sulfate, 5 days)
Other: standard of care (SOC) for COVID-19 — Standard of care (SOC) for COVID-19
  Arms: Second Arm (Continued Standard of Care (SOC) Therapy)

SUMMARY:
This is a pilot, randomized, single-center, parallel group, open-label controlled study to evaluate the feasibility, safety, efficacy, and pharmacokinetics of nebulized HCQ01 plus Standard of Care (SOC) versus SOC alone in hospitalized COVID-19 patients. The Jordanian Ministry of Health (MOH) is the study sponsor, and the study will be conducted at MOH COVID-19 hospitals.

Approximately 110 patients, ≥18 years of age with a confirmed SARS-CoV-2 infection, will be enrolled and randomized 1:1 to the treatment and control arms where they will receive ten doses of Hydroxychloroquine solution via nebulizer in addition to SOC or the control arm where treatment will follow the MOH SOC.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant (positive β-human chorionic gonadotropin test, β-HCG) or lactating female at screening.
2. Patients with a history of retinopathy, sickle cell disease or trait, psoriasis, porphyria, history of splenectomy, mental illness or uncontrolled seizures disorder, known active tuberculosis or history of incompletely treated tuberculosis, patients on chronic immunosuppression for other medical conditions such as rheumatological disorders, inflammatory bowel disease, or in patients with organ transplants.
3. Patients admitted in ICU.
4. Taking medications which may lead to interactions with hydroxychloroquine, including penicillamine, telbivudine, botulinum toxin, fluconazole, digoxin, propafenone , cimetidine, statins, warfarin, and cyclosporine within 2 weeks of dosing start, and during the duration of the study.
5. History of Glucose-6-phosphate dehydrogenase deficiency.
6. Pre-treatment corrected QT interval (QTc) ≥450 milliseconds.

Exclusion Criteria:

1. Pregnant (positive β-human chorionic gonadotropin test, β-HCG) or lactating female at screening.
2. Patients with a history of retinopathy, sickle cell disease or trait, psoriasis, porphyria, history of splenectomy, mental illness or uncontrolled seizures disorder, known active tuberculosis or history of incompletely treated tuberculosis, patients on chronic immunosuppression for other medical conditions such as rheumatological disorders, inflammatory bowel disease, or in patients with organ transplants.
3. Patients admitted in ICU.
4. Taking medications which may lead to interactions with hydroxychloroquine, including penicillamine, telbivudine, botulinum toxin, fluconazole, digoxin, propafenone , cimetidine, statins, warfarin, and cyclosporine within 2 weeks of dosing start, and during the duration of the study.
5. History of Glucose-6-phosphate dehydrogenase deficiency.
6. Pre-treatment corrected QT interval (QTc) ≥450 milliseconds.
7. Acute or chronic kidney disease (stage-4 or -5 renal impairment; eGFR<30 mL/min/1.73 m2 or hemodialysis).
8. Liver Child-Pugh grade C.
9. Patients with Hypokalemia (<3.5mmol/L), Hypocalcemia (<2.2mmol/L), Hypomagnesemia (<0.66mmol/L). Will be included after correction.
10. Need for mechanical ventilation.
11. History of hypersensitivity to hydroxychloroquine.
12. History of Chronic Hepatitis B or hepatitis C infections.
13. History of Human Immunodeficiency Virus (HIV) infection.
14. Concurrent serious illness including, but not limited to, any of the following:

    * Clinically significant cardiovascular disease (e.g., uncontrolled hypertension, myocardial infarction, or unstable angina).
    * New York Heart Association class II-IV congestive heart failure.
    * Serious cardiac arrhythmia requiring medication. -Peripheral vascular disease ≥ grade 2 within the past year. -
    * Psychiatric illness/social situation that would limit compliance with study requirements. -COPD, Lung cancer, and moderate to severe asthma.
15. Any other significant finding based on the judgment of the PI would increase the risk of having an adverse outcome from participating in this study.
16. Any other concomitant treatment based on the judgment of the PI would increase the risk of having an adverse outcome from participating in this study.
17. Is currently participating in or has participated in an interventional clinical trial with an investigational compound or device within 80 days of signing the informed consent/assent for this current trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-03-20 (Estimated); Primary Completion 2022-07-20 (Estimated); Study Completion 2022-07-20 (Estimated)

PRIMARY OUTCOMES:
WHO Ordinal Scale for for Clinical Improvement | [ Day -1 (screening) to Days 3,6, and 14 ]
  Change in condition measured using the Ordinal Scale for Clinical Improvement. Patients are scored on a scale of 0-10 with 0 being uninfected and 10 being dead

SECONDARY OUTCOMES:
Proportion of participants who improve by at least one level lower on the 11-point WHO-OSCI | Day 28
All-cause mortality | Day 28
HCQ concentration in plasma versus time profiles | Day 1 pre-dose (within 1-hour prior dosing) and +2, +5, +10, +15, +20, +25, and +30 minutes after dose, and also +1, +2, +3, +4 and +6 hours post-dose completion
Change from Baseline Oxygenation as determined by the SpO2/FiO2 ratio | Days 3 & 6
Rate of Transfer to the Intensive Care Unit | Up to day 28
Time to Hospital Discharge or NEWS2 (National Early Warning Score 2) of ≤ 2 | Up to day 28
Treatment-related adverse events of HCQ | Up to day 28
Cardiac Arrhythmia - Polymorphic Ventricular Tachycardia [Time Frame | Up to day 6
  Cardiologist Diagnostic Documentation
Cardiac Arrhythmia - Ventricular Tachycardia | Up to day 6
  Cardiologist Diagnostic Documentation
Cardiac Arrhythmia - Lengthening QTc | Up to day 6
  Cardiologist Diagnostic Documentation

CONTACTS AND LOCATIONS:
Overall Officials: Feras Hawari, MD, Principal Investigator — The Jordanian Ministry of Health
Locations (1):
- Prince Hamza Hospital/ Amman Field Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No